CLINICAL TRIAL: NCT02189811
Title: Polio End-game Strategies - Poliovirus Type 2 Challenge Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ali Faisal Saleem, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEGS
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Poliomyelitis
Keywords: IPV; OPV; tOPV; bOPV; Polio; Endgame; Pakistan
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- IPV (Experimental): IPV at birth, 6 weeks, 10 weeks, 14 weeks, followed by tOPV at 18 and 22 weeks
  Interventions: Biological: IPV
- bOPV (Experimental): bOPV at birth, 6, 10, and 14 weeks. followed by tOPV at 18 and 22 weeks of age
  Interventions: Biological: bOPV
- bOPV and IPV (Experimental): bOPV at birth, 6, 10 weeks, and IPV+bOPV at 14 weeks, and tOPV at 18 and 22 weeks of age
  Interventions: Biological: bOPV and IPV
- bOPV and IPV and IPV2 (Experimental): bOPV at birth, 6, 10 weeks and bOPV+IPV at 14 weeks and tOPV+IPV2 at 18 weeks and tOPV alone at 22 weeks of age
  Interventions: Biological: bOPV and IPV and IPV2
- tOPV (Active Comparator): tOPV at birth, 6, 10, 14, 18 and 22 weeks of age
  Interventions: Biological: tOPV

INTERVENTIONS:
Biological: IPV — IPV at birth, 6, 10, 14 weeks of age and tOPV at 18 and 22 weeks of age
  Arms: IPV
Biological: bOPV — bOPV at birth, 6, 10, 14 weeks and tOPV at 18 and 22 weeks of age
  Arms: bOPV
Biological: bOPV and IPV — bOPV till week 10, bOPV+IPV at 14 and tOPV at 18 and 22 weeks of age
  Arms: bOPV and IPV
Biological: bOPV and IPV and IPV2 — bOPV till week 10, bOPV+IPV at 14, tOPV+IPV2 at 18 and tOPV at 22 weeks of age
  Arms: bOPV and IPV and IPV2
Biological: tOPV — tOPV till 22 weeks of age
  Arms: tOPV

SUMMARY:
Poliomyelitis eradication has entered its last phase with only three remaining endemic countries, of which Pakistan is one. There hasn't been a case of wild type poliovirus 2 since 1999, and no case of wild type poliovirus 3 since November 2012. However, paralytic polio resulting from circulating strains of Sabin poliovirus type 2 have become a challenge, and reported from several areas with low population immunity to polio, including in Pakistan. This study will provide data to National Immunization Authorities in order to make strategic decisions about their polio vaccination schedules in anticipation of the global tOPV to bOPV switch and will provide data on the proposed responses to type 2 poliovirus outbreaks.

DETAILED DESCRIPTION:
The "Polio Endgame Strategy" consists of set of tasks and activities that will be implemented in the next five years. It includes gradual withdrawal of the widely used oral poliomyelitis vaccine (OPV) containing live poliovirus, and will eventually lead to complete eradication and containment of all wild, vaccine-related (VDPV) and Sabin polioviruses. The withdrawal of the type 2 components of trivalent OPV (tOPV) is the key component in the elimination of cVDPVs. This entails strengthening of the immunization system by introducing at least one dose of affordable IPV into the routine immunization schedule globally and then replacing the trivalent OPV with bivalent OPV in all OPV-using countries - setting the stage for eventually ending bOPV use in 2019-2020. Most of the developing countries have an OPV schedule however many developed and European countries follow the IPV only schedule. The current recommendations for polio eradication and endgame is IPV vaccine to be administered together with third OPV dose, which in most countries occurs at 14 weeks of age.

This study will assess the protection to type 2 poliovirus achieved after completion of the recommended schedule with bOPV and IPV; it will compare immunogenicity of bOPV + IPV schedule with tOPV only schedule; and will quantify the cross-reactivity of bOPV on inducing type 2 immunological reaction. In addition, it will also provide first data on the proposed outbreak response to type 2 (either with mOPV 2 or with a combination of mOPV 2 and IPV 2).

This study will provide data to National Immunization Authorities in order to make strategic decisions about their polio vaccination schedules in anticipation of the global tOPV to bOPV switch and will provide data on the proposed responses to type 2 poliovirus outbreaks.

ELIGIBILITY:
Inclusion Criteria:

* Newborn of either gender born healthy with birth weight 2.0 kg or more, with immediate cry, at the study sites (home or health facility births)
* Not planning to travel away during entire the study period (birth-154 days; birth 22 weeks).
* Parents resident of the study area for last 3 month at the time of enrolment
* Parent/guardian provides informed consent

Exclusion Criteria:

* Newborns found acutely ill at the time of enrolment and requiring emergent medical care/hospitalization, birth weight below 2.0 kg, cry >2 minutes after birth, or family is planning to be absent during the birth - 154 days study period
* Refusal of blood testing and cord blood testing
* Receipt of OPV after birth before eligibility screen
* Newborns with certain medical conditions i.e., syndromic infants, neonate with petechial or purpura (contraindication of intramuscular injections)
* A diagnosis or suspicion of immunodeficiency disorder (either in the participant or in a member of the immediate family - e.g. several early infant deaths, household member on chemotherapy) will render the newborn ineligible for the study.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in seroprevalence of neutralizing antibodies for type 2 in 19 weeks of age between arms | 19 weeks of age

SECONDARY OUTCOMES:
Seroprevalence of neutralizing antibodies at 18 weeks of age | 18 weeks of age

OTHER OUTCOMES:
Difference in shedding of poliovirus type 2 in stool in 19 weeks of age between arms | 19 weeks of age
Difference in seroprevalence of neutralizing antibodies at 22 weeks of age between arms | 22 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Saleem, MBBS,FCPS,MSc, Principal Investigator — Aga Khan University
Locations (1):
- Rehri goth, Ibrahim Hyderi, Ali Akbar Shah, and Bhens Colony, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Saleem AF, Yousafzai MT, Mach O, Khan A, Quadri F, Weldon WC, Oberste MS, Zaidi SS, Alam MM, Sutter RW, Zaidi AKM. Evaluation of vaccine derived poliovirus type 2 outbreak response options: A randomized controlled trial, Karachi, Pakistan. Vaccine. 2018 Mar 20;36(13):1766-1771. doi: 10.1016/j.vaccine.2018.02.051. Epub 2018 Feb 21. PMID 29477307